CLINICAL TRIAL: NCT01976117
Title: E-nose Utility in the Diagnosis of Bacterial Infection in Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: E-nose Utility in the Diagnosis of Bacterial Infection in COPD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: IIBSP-ENO-2009-21
Record Dates: First submitted 2013-10-22; First posted 2013-11-05 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-09

CONDITIONS: Pulmonary Disease, Chronic Obstructive (COPD)
MeSH Terms: conditions — Lung Diseases; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- enose (Experimental)
  Interventions: Device: enose

INTERVENTIONS:
Device: enose

SUMMARY:
Hypothesis: A commercial e-nose (Cyranose 320) is able to detect specific breathprints from patients with COPD and bacterial infection

DETAILED DESCRIPTION:
Thirty to 50% of COPD patients have airway colonization with potentially pathogenic bacteria. This is associated with worse prognosis. Currently, diagnosis of bacterial colonization relies mainly upon quantitative sputum culture. However, this method lacks good sensitivity. The electronic nose is a novel device made up of nanosensors capable of detecting specific volatile organic compounds (VOCs). OBJECTIVES: Main 1) To assess the usefulness of the electronic nose in the diagnosis of bacterial colonization in COPD. Secondary 1) To define the VOCs pattern associated with bacterial colonization. 2) To study the pattern of pulmonary and systemic inflammation associated with bacterial colonization as well its relationship with the aforementioned VOCs patterns.

ELIGIBILITY:
Inclusion Criteria:

* COPD patients

Exclusion Criteria:

* Exacerbation in the last 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2012-06; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Breathprint in exhaled breath from patients with COPD | Day 1
  Breathprints will be assessed by discriminant analysis on principal component reduction, resulting in cross-validated accuracy values

SECONDARY OUTCOMES:
Breathprint in exhaled breath from COPD patients with bacterial colonization | Day 1
  Breathprints will be assessed by discriminant analysis on principal component reduction, resulting in cross-validated accuracy values

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona, Spain

REFERENCES:
- [Derived] Sibila O, Garcia-Bellmunt L, Giner J, Rodrigo-Troyano A, Suarez-Cuartin G, Torrego A, Castillo D, Solanes I, Mateus EF, Vidal S, Sanchez-Reus F, Sala E, Cosio BG, Restrepo MI, Anzueto A, Chalmers JD, Plaza V. Airway Mucin 2 Is Decreased in Patients with Severe Chronic Obstructive Pulmonary Disease with Bacterial Colonization. Ann Am Thorac Soc. 2016 May;13(5):636-42. doi: 10.1513/AnnalsATS.201512-797OC. PMID 26882402